CLINICAL TRIAL: NCT06417710
Title: Standardized Clinical Assessment of Patients With Leptomeningeal Metastasis
Acronym: NANO-LM
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: M.D. Anderson Cancer Center (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NANO-LM-01
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Leptomeningeal Metastasis; Leptomeningeal Disease; Leptomeningeal Neoplasms; Leptomeningeal Cancer
MeSH Terms: conditions — Meningeal Carcinomatosis; Meningeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neurological Assessment — Clinical neurological assessment performed by 2 raters

SUMMARY:
The goal of this project is to develop and validate a reproducible scorecard for the neurological assessment of patients with leptomeningeal metastases that can be used in clinical trials including such patients, as well as in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or more), female or male
* Histologically confirmed diagnosis of extra-CNS primary solid cancer
* Diagnosis of leptomeningeal metastases confirmed or probable per EANO ESMO criteria
* Performance status compatible with enrolment into clinical trials
* Ability to consent
* Signed informed consent form from patient
* Participation in a parallel clinical trial is allowed in this non-interventional study

Exclusion Criteria:

* Inability to give informed consent
* Inability to adhere to recommended follow-up according to the treating physician

Vulnerable participants will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with leptomeningeal metastases from various extra-central nervous system (CNS) solid primary tumors for whom a tumor-specific treatment is planned
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
inter-observer agreement of response assessment of the overall clinical assessment - per center and among all raters | December 2026

SECONDARY OUTCOMES:
inter-observer reproducibility (agreement) for each item - per center and among all raters | December 2026
association between items | December 2026
variability of the interobserver agreement | December 2026
description of clinical neurological symptoms and signs | December 2026
association of clinical response with imaging and CSF cytology response and the overall global clinical/MRI/CSF response | December 2026

CONTACTS AND LOCATIONS:
Locations (3):
- MD Anderson Cancer Center, Houston, Texas, United States
- Netherlands Cancer Institute, Amsterdam, Netherlands
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Le Rhun E, Nayak L, Lim-Fat MJ, Ruda R, Pentsova E, Forsyth P, O'Brien BJ, Preusser M, Kumthekar P, Brandsma D, Weller M. NANO-LM: An updated scorecard for the clinical assessment of patients with leptomeningeal metastases. Neuro Oncol. 2025 Feb 10;27(2):455-465. doi: 10.1093/neuonc/noae171. PMID 39208403